CLINICAL TRIAL: NCT00290277
Title: Evaluate the Immunogenicity & Safety of GSK Biologicals' HPV-16/18 L1/AS04 Vaccine Administered Intramuscularly According to a 0,1,6 Mth Schedule in Healthy Female Subjects Aged 10-14 Yrs
Brief Title: Evaluate the Immunogenicity & Safety of GSK Biologicals' HPV Vaccine in Female Subjects Aged 10-14 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 104951
Record Dates: First submitted 2006-02-10; First posted 2006-02-13 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Infections, Papillomavirus
MeSH Terms: conditions — Papillomavirus Infections

INTERVENTIONS:
Biological: HPV-16/18 L1/AS04

SUMMARY:
Human papillomavirus infection has clearly been recognized as the cause of cervical cancer. Indeed, the infection of the cervix by certain oncogenic types of HPV, if not cleared , can lead over time to cervical cancer in women . This study will evaluate the immunogenicity and the safety of the HPV vaccine in female subjects aged 10 - 14 years in Korea.

DETAILED DESCRIPTION:
Study participants will receive either HPV or hepatitis A vaccine, study duration will last for 7 months and involve a total of 4 visits.

ELIGIBILITY:
Inclusion criteria:

* A female subject between, and including, 10 and 14 years of age at the time of the first vaccination.
* Written informed assent from the subject and informed consent from the parent or guardian of the subject should be obtained prior to enrolment.
* Subjects must have a negative urine pregnancy test.
* Healthy subject before entering the study as established by medical history and clinical examination.
* Subject must be of non-childbearing potential.

Exclusion criteria:

* Pregnant or breastfeeding.
* Previous vaccination against HPV.
* Known acute or chronic, clinically significant neurologic, hepatic or renal functional abnormality
* History of chronic condition(s) requiring treatment such as cancer, chronic hepatic or kidney disease(s), diabetes, or autoimmune disease."

Ages: 10 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2005-11; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
To evaluate antibody responses against HPV-16 and HPV-18 in all HPV vaccine recipients at Month 7.

SECONDARY OUTCOMES:
To evaluate safety and reactogenicity throughout the study period.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- South Korea (3):
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Kwangju
  - GSK Investigational Site, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 104951 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 104951 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 104951 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 104951 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 104951 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 104951 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 104951 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register